CLINICAL TRIAL: NCT00509249
Title: A Phase II Study of VEGF Trap (NSC 724770) in Patients With MDS
Brief Title: Aflibercept in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination for discouraging results
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00180; PHII-73; N01CM62209 (NIH); CDR0000558101 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2012-11

CONDITIONS: Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients will receive aflibercept IV at 4 mg/kg over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well aflibercept works in treating patients with myelodysplastic syndromes. Aflibercept may be able to carry cancer-killing substances directly to myelodysplastic syndrome cells. It may also stop the growth of cancer cells by blocking blood flow to the cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the antitumor activity of aflibercept as assessed by the hematological response rate.

II. To determine overall and progression-free survival in patients with myelodysplastic syndromes.

III. To assess hematologic improvement and time to leukemic transformation. IV. To assess the toxicity profile of aflibercept in this patient population. V. To perform correlative studies to better understand the ability of aflibercept to reach and modulate its respective targets.

OUTLINE: This is a multicenter study.

Patients will receive aflibercept IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples will be obtained periodically for pharmacokinetic and biomarker correlative studies. Pharmacokinetic analysis by ELISA; anti-aflibercept antibody measurements; analysis of VEGF and VEGFR expression; and analysis of gene expression by quantitative PCR will be conducted. The effect of aflibercept on apoptosis and proliferation of CD34+ cells will also be analyzed by flow cytometry based assays.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed myelodysplastic syndromes (MDS), including any of the following:

  * Secondary MDS
  * MDS/myeloproliferative disorders (MPD) (e.g., chronic myelomonocytic leukemia or atypical chronic myeloid leukemia)
  * IPSS scores of 0.5 or greater (≥ INT-1) OR transfusion dependent despite use of growth factors
  * No more than 20% blasts in the marrow
  * Patients who have not responded after 3 courses of hypomethylating agents (azacitidine or decitabine) OR; who are unable to tolerate hypomethylating agents OR who refused to receive hypomethylating agents are eligible for this study
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST/ALT ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio < 1 OR urine protein < 500 mg by 24-hour urine collection
* PT INR ≤ 1.5
* Patients with PT INR > 1.5 on full-dose anticoagulants (e.g., warfarin) are eligible provided both of the following criteria are met:

  * Patient has an in-range INR (usually between 2 and 3) and is on a stable dose of oral anticoagulant or low molecular weight heparin
  * Patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 6 months after completion of study treatment
* Prior DNA-demethylating agent therapy or lenalidomide therapy allowed
* Prior treatment with other molecular agents, such as thalidomide, valproic acid, or imatinib mesylate allowed

Exclusion Criteria:

* Evidence of active malignancies other than squamous cell or basal cell carcinoma of the skin
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study
* Serious or non-healing wound, ulcer, or bone fracture
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* Significant traumatic injury within the past 28 days
* Clinically significant cardiovascular disease, including any of the following:

  * History of cerebrovascular accident (CVA) within the past 6 months
  * Uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg or systolic BP > 180 mm Hg if diastolic blood pressure < 90 mm Hg (on at least 2 repeated determinations on separate days) within the past 3 months
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class III or IV congestive heart failure, serious cardiac arrhythmia requiring medication, or unstable angina pectoris within the past 6 months
* Clinically significant peripheral vascular disease within the past 6 months
* Pulmonary embolism, deep vein thrombosis (DVT), or other thromboembolic event within the past 6 months
* Evidence of bleeding diathesis or coagulopathy
* Concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situation that would limit compliance with study requirements
* Prior cytotoxic chemotherapy for MDS
* Molecular therapy or immunosuppressive agents (including steroids) within the past 3 weeks
* Other prior antiangiogenesis agents
* Coronary artery bypass graft (CABG) within the past 6 months
* Valproic acid should be discontinued at least 24 hours before aflibercept administration, unless needed for seizure control
* Major surgical procedure or open biopsy within the past 28 days
* Core biopsy (other than bone marrow biopsy) within the past 7 days
* Anticipation of need for major surgical procedures during the course of the study
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 71 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Hematological Response Rate
Description: Complete Response (CR): repeat bone marrow (BM) shows <5% myeloblasts, and peripheral blood values lasting ≥ 2 months of hemoglobin (hgb) (>110 g/L), neutrophils (≥1.0x10^9/L), platelets (≥100x10^9/L), blasts (0%) and no dysplasia. Partial Response (PR): same as CR for peripheral blood except BM shows blasts decrease by ≥ 50% but still > 5% or a less advanced FAB classification from pretreatment. Hematological response=CR+PR.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Description: "Other" Adverse Events table includes events of all grades and attributions to treatment not included in the "Serious" Adverse Event table.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (107)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (2)
Cardiac disorder (Cardiac disorders) | 1 (4)
Cardiac pain (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (7)
Flashing vision (Eye disorders) | 1 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 5 (20)
Diarrhea (Gastrointestinal disorders) | 5 (14)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (6)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (12)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Toothache (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 3 (8)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 4 (9)
Disease progression (General disorders) | 3 (3)
Edema limbs (General disorders) | 6 (33)
Fatigue (General disorders) | 12 (36)
Fever (General disorders) | 3 (4)
Flu-like symptoms (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Abdominal infection (Infections and infestations) | 1 (5)
Gingival infection (Infections and infestations) | 1 (2)
Joint infection (Infections and infestations) | 1 (3)
Opportunistic infection (Infections and infestations) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Vaginal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (17)
Fracture (Injury, poisoning and procedural complications) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (14)
Alkaline phosphatase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 8 (19)
Bilirubin increased (Investigations) | 3 (7)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (17)
Electrocardiogram QTc interval prolonged (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 8 (52)
Lymphocyte count decreased (Investigations) | 4 (20)
Neutrophil count decreased (Investigations) | 9 (51)
Platelet count decreased (Investigations) | 11 (74)
Weight loss (Investigations) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 5 (10)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (13)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (12)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (15)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (18)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (13)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Ataxia (Nervous system disorders) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (18)
Headache (Nervous system disorders) | 9 (30)
Neurological disorder NOS (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4)
Seizure (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (8)
Taste alteration (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (12)
Insomnia (Psychiatric disorders) | 2 (6)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (2)
Protein urine positive (Renal and urinary disorders) | 5 (16)
Urinary frequency (Renal and urinary disorders) | 2 (15)
Urinary incontinence (Renal and urinary disorders) | 2 (5)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (22)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (55)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (4)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 5 (17)
Sweating (Skin and subcutaneous tissue disorders) | 3 (17)
Hematoma (Vascular disorders) | 2 (15)
Hypertension (Vascular disorders) | 8 (44)
Lymphedema (Vascular disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Study was terminiated after completion of the first stage due to a lack of activity (no hematological responses were observed).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less